CLINICAL TRIAL: NCT05775796
Title: A Single-arm, Multicenter, and Phase II Clinical Study to Evaluate the Efficacy and Safety of Serplulimab Combined With Chemotherapy in Neoadjuvant and Adjuvant Treatment of Resectable Stage II-IIIA NSCLC
Brief Title: Evaluate the Efficacy and Safety of Serplulimab Plus Chemotherapy in Neoadjuvant and Adjuvant Treatment of Resectable NSCLC (ECTOP-1013)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haiquan Chen, Director of Thoracic Surgery, Fudan University Shanghai Cancer Center, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX10IIT21
Record Dates: First submitted 2023-03-07; First posted 2023-03-20 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Non-small Cell Lung Cancer; Stage II-IIIA; Immunotherapy; Neoadjuvant Therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Serplulimab plus platinum doublet chemotherapy (Experimental)
  Interventions: Drug: Serplulimab and Chemotherapy

INTERVENTIONS:
Drug: Serplulimab and Chemotherapy — Serplulimab+Paclitaxel+Cisplatin/Carboplatin Serplulimab+Pemetrexed+Cisplatin/Carboplatin

SUMMARY:
This is a clinical trial from Eastern Cooperative Thoracic Oncology Project (ECTOP), numbered as ECTOP-1013. The purpose of this neoadjuvant and adjuvant study is to evaluate the efficacy and safety of Serplulimab and chemotherapy in treating resectable Non-Small Cell Lung Cancer(NSCLC). The study also intended to explore the immune function of tumor-draining lymph nodes during immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* stage IB-IIIA, operable non-small cell lung cancer, confirmed in tissue.
* Able and willing to give written informed consent and has signed the informed consent form (ICF), prior to performance of any trial activities.
* Eligible male and female subjects aged 18-75 years.
* Lung function capacity capable of tolerating the proposed lung surgery.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.
* Available tissue of primary lung tumor.

Exclusion Criteria:

* Presence of locally advanced, inoperable or metastatic disease.
* Subjects with EGFR mutation or ALK、ROS1 gene rearrangement.
* Active, known or suspected autoimmune disease.
* Prior treatment with any drug that targets T cell co-stimulations pathways (such as checkpoint inhibitors).

Other protocol defined inclusion/exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Rate of Major Pathologic Response (MPR) | Up to 6 months
  Major pathologic response (MPR) rate is defined as after neoadjuvant treatment, the percentage of residual tumor cells in the tumor bed ≤ 10%, regardless of the proportion of patients with residual tumor cells in lymph nodes

SECONDARY OUTCOMES:
Rate of Pathologic Complete Response (pCR) | Up to 6 months
  Proportion of patients without residual tumor cells in tumor bed and lymph nodes after neoadjuvant therapy
Rate of R0 resection | Up to 6 months
  The complete resection rate is the proportion of patients with complete resection
Objective remission rate(ORR) | Up to 6 months
  Objective response rate according to RECIST 1.1
Event-Free Survival (EFS) | 2 years
  Event-free survival (EFS) is defined as the length of time from enrollment to any of the following events: any progression of disease precluding surgery, progression or recurrence disease assessment per response evaluation criteria in solid tumors (RECIST) 1.1 after surgery, or death due to any cause. Patients who don't undergo surgery for reason other than progression will be considered to have an event at progression or death.
Immune infiltrations in tumor-draining lymph nodes | 2 years
  Immune cell subtype infiltrations in tumor-draining lymph nodes by single-cell sequencing

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No